CLINICAL TRIAL: NCT00927537
Title: Data Collection on Hypertension and Its Treatment With Kinzal®/ Kinzalplus®
Brief Title: Therapy of Essential Hypertension With Kinzal®/ Kinzalplus®
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13599; KL0810CH (Other: company internal)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Hydrochlorothiazide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Drug: Telmisartan (Kinzal/Pritor, BAY68-9291)
- Group 2
  Interventions: Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) + Hydrochlorothiazide

INTERVENTIONS:
Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) — Patients under daily life treatment receiving Kinzal according to local drug information.
  Groups: Group 1
Drug: Telmisartan (Kinzal/Pritor, BAY68-9291) + Hydrochlorothiazide — Patients under daily life treatment receiving Kinzalplus according to local drug information.
  Groups: Group 2

SUMMARY:
The efficacy and tolerability of an antihypertensive treatment with Telmisartan is followed over 3-4 months

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients seen by the physician requiring antihypertensive treatment

Exclusion Criteria:

* According to the local drug information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 2052 (Actual)
Dates: Start 2008-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Blood pressure | After 1-2 weeks, 1month, 3-4 months

SECONDARY OUTCOMES:
Change in Mean heart rate (bpm) | Baseline and 3-4 month
Change in Mean Weight (kg) | Baseline and 3-4 month
Change in Mean laboratory parameters (total cholesterol, LDL, HDL, triglyceride, fasting blood glucose) | Baseline and 3-4 month
Patient Medical History: Duration of hypertension, Pre-treatment of hypertension, Comorbidities and Concomitant treatment | Baseline
Final evaluation of efficacy (very good, good, sufficient, insufficient) and tolerability (very good, good, sufficient, insufficient) of treatment by the physician. | After 3-4 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Switzerland